CLINICAL TRIAL: NCT01469312
Title: Effect of Pasta on Blood Glucose Response in Normal Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Minneapolis Veterans Affairs Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Frank Q. Nuttall, MD, PhD, Chief, Section of Endocrinology, Metabolism & Nutrition, Professor of Medicine, Minneapolis Veterans Affairs Medical Center
Allocation: Randomized | Model: Crossover | Masking: Single
Other Study IDs: 4231
Record Dates: First submitted 2011-11-03; First posted 2011-11-10 (Estimated); Last update posted 2011-11-11 (Estimated); Status verified 2011-11

CONDITIONS: Blood Glucose Concentration; Type 2 Diabetes; Metabolic Syndrome
Keywords: Low Biologically Available Glucose Diet (LoBAG diet); Diabetes; Glycemic Index
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Metabolic Syndrome; Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Placebo Comparator): The control arm consists of the traditional pasta.
  Interventions: Other: modified pasta
- Modified pasta (Active Comparator): Dreamfields, Miracle Noodles
  Interventions: Other: modified pasta

INTERVENTIONS:
Other: modified pasta — 50 grams carbohydrate as a single breakfast meal
  Other Names: Dreamfields Pasta, Miracle Noodles

SUMMARY:
The objective of this study is to determine whether ingestion of modified pasta products (Dreamfields, Miracle Noodles) result in an improvement in blood glucose concentration when compared with a traditional pasta.

DETAILED DESCRIPTION:
On one occasion the pasta will be a traditionally available pasta; on another occasion, approximately 1 week later a modified pasta, advertised to contain ~ 5 grams of digestible carbohydrate, or to be low in digestible starch, will be studied.

ELIGIBILITY:
Inclusion Criteria:

* Normal blood glucose concentration

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2010-04; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Change in Blood Glucose | 0, 30, 60, 90, 120, and 180 minutes after ingestion
  Blood glucose will be determined by finger stick.

CONTACTS AND LOCATIONS:
Overall Officials: Frank Q Nuttall, M.D., Ph.D., Principal Investigator — Minneapolis Veterans Affairs Medical Center; Mary C Gannon, Ph.D., Principal Investigator — Minneapolis Veterans Affairs Medical Center
Locations (1):
- Minneapolis VA Health Care System, Minneapolis, Minnesota, United States

REFERENCES:
- [Background] Nuttall FQ, Schweim K, Hoover H, Gannon MC. Effect of the LoBAG30 diet on blood glucose control in people with type 2 diabetes. Br J Nutr. 2008 Mar;99(3):511-9. doi: 10.1017/S0007114507819155. Epub 2007 Sep 10. PMID 17868489